CLINICAL TRIAL: NCT06781047
Title: Serebral Palsili Adölesanlarda Gövde Odaklı Rehabilitasyonun Spinal Mobilite, Gövde Kontrolü ve El Fonksiyonları Üzerine Etkilerinin İncelenmesi
Brief Title: Effects of Trunk-Focused Rehabilitation on Spinal Mobility, Trunk Control, and Hand Functions in Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Saglik Bilimleri U, 26848; 0000-0002-4321-2332 (Registry Identifier: Gül EVDALI); 0000-0001-9120-7071 (Registry Identifier: Seval KUTLUTÜRK YIKILMAZ)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy (CP); Adolescent; Trunk; Exercise
Keywords: cerebral palsy, trunk training, trunk control exercise
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trunk Focused Rehabilitation (TFR) plus Conventional Rehabilitation (CR) Group (Experimental): 1. Abdominal stabilization progression for TFR is applied to all cases with simultaneous breathing exercises for 8 weeks (24 sessions in total) (8). Exercises are performed 3 days a week, 45 minutes a day, starting from warm-up and recumbent position respectively, and the intensity is adjusted individually by observing tone and motivation.
  The experimental group's routine physiotherapists also gave them a conventional rehabilitation program (the same protocol as in the active comparison arm) for 40 minutes per day, 2 days per week.
  Interventions: Other: Trunk Focused Rehabilitation (TFR); Other: Conventional Rehabilitation (CR)
- Conventional Rehabilitation (CR) Group (Active Comparator): The control group is the group that receives conventional treatment 2 days a week, 40 minutes per session.
  Conventional Rehabilitation Program Content: All sessions include the following rehabilitation program, supervised by a physiotherapist and individualized according to tolerance. Number of exercise repetitions: 10-20. The intensity is adjusted by observing motivation.
  Interventions: Other: Conventional Rehabilitation (CR)

INTERVENTIONS:
Other: Trunk Focused Rehabilitation (TFR) — Abdominal stabilization progression for TFR is applied with simultaneous breathing exercise for 3 days a week, 45 minutes a day, 8 weeks (24 sessions in total)(8).
  1. Basic Abdominal Stabilization Training, Task-Focused Exercises (without spinal diagonal and rotational components)(8,12).
     Warm-up: 5 minutes, Global Stretching and Relaxation(9,10,11). Extremity load, elastic band, and unstable surface are added as stabilization is achieved in neurodevelopmental positions. Task-oriented exercises(12).
     Cooling Down: Warm-up exercises are repeated.
  2. General Posture and Asymmetry Training Brochure (includes adolescent, family, and team members)(13-17).
  The exercise starts with 3 seconds and gradually progresses to 10 seconds, 10 repetitions, and 3 sets.
  The TFR group also receives Conventional Treatment 2 days a week, 40 minutes per day, for 8 weeks. The same treatment protocol is applied as the control group). Routine physiotherapists apply conventional treatment.
  Arms: Trunk Focused Rehabilitation (TFR) plus Conventional Rehabilitation (CR) Group
Other: Conventional Rehabilitation (CR) — Conventional treatment is applied to the group, 2 days a week, 40 minutes each session, for 8 weeks. It is an intervention performed by a physiotherapist who regularly follows up in a special education and rehabilitation center.
  1. Normal Joint Movement (NEH)
  2. Stretching for the lower, and upper extremities and around the hips
  3. Lying activities
  4. Curl up (assisted, unaided)
  5. Bridging exercise, cat camel exercise, posterior pelvic tilt exercise
  6. Walking training
  7. Climbing and descending stairs
  8. Weight transfer exercises at standing, sitting

SUMMARY:
Main Purpose: This study aims to investigate the effects of trunk-focused rehabilitation on trunk control, spinal mobility, and manual skills in adolescents with cerebral palsy (CP).

Secondary Purpose: To investigate its effects on functional health.

DETAILED DESCRIPTION:
Muscle weakness in the trunk; reducing the support of children with CP, may cause increased distal tone and decreased function in their daily practices. When the effectiveness of interventions that can improve postural control is evaluated, trunk-focused training is one of the 5 interventions supported by a moderate level of evidence. In an intervention study where trunk training was structured individually, there may be an improvement in erector spinae muscle group scores when evaluated with sEMG. A study of 28 cases, including all subtypes of CP, aimed to evaluate the inter-rater reliability of Spinal Mouse (SM) and the effect on the spinal column with 4 hours a day, 1 week of intensive clinical rehabilitation application. In this population, SM was evaluated with therapeutic interventions, it has been reported that it may show significant posture differences, especially in total spinal inclination and spine length. In children aged 5-12 years with Gross Motor Function Classification System (GMFCS) Level 1, 2 CP, there are significant improvements in the Trunk Control Measurement Scale (TCMS) score after only Trunk Focused Rehabilitation (TFR). It is emphasized that with TFR, which is described as a unique approach, postural control of the whole body can be improved by the use of intermediate postures and postural activities involving the trunk and better participation of the affected muscles. Only after TFR intervention, the findings of improvement in the assessments on a 3D force platform were highlighted in postural sway, early sternal and sacral decelerations. It is carried out with active participation, individualized, intensive, and time-limited, considering possible content limitations and the needs and preferences of the adolescent and the family. It is stated that trunk-targeted interventions can be given together with conventional physical therapy programs to support functional improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Levels 1 and 2 according to Gross Motor Function Classification System (GMFCS)
2. Viking Speech Scale Turkish version/(VSS-T) 1-2 level, understood to speak and able to take commands
3. Adolescents with CP between the ages of 12-18
4. Those whose guardian / legal representative and themselves have received an Informed Voluntary Consent Form
5. No hip dislocation
6. Scoliosis below 25 degrees according to the radiographic evaluation made in the last 6 months

Exclusion Criteria:

1. Having had any surgery related to the intrathecal baclofen pump
2. Having botulinum toxin injection treatment or orthopedic surgery within the last 6 months
3. Having severe vision, hearing, and cognitive deficiencies
4. Acute medical illness

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Trunk Control | at baseline and week 9
  Trunk Impairment Scale: It consists of coordination, dynamic and static sections. In the static section, the responses in actively and passively crossing the legs with the feet in a supported position are recorded. In the dynamic section, unilateral hip movements and lateral flexion of the trunk are evaluated. In the coordination section, the upper and lower body are asked to move. Coordination consists of dynamic and static sections. The maximum scores that can be obtained from the tests are 7 for the static section, 10 for the dynamic section, and 6 for the coordination section. The score range is 0-23. The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance.
Evaluation of Spinal Mobility | at baseline and week 12
  Spinal Mobility and Alignment Assessment (Sagittal Plane): Spinal Mouse (SM) measurements are taken at the same time of day, in an environment where the patient is resting, distrubating their weight equally between their two feet as much as possible, and standing symmetrically, while the patient is standing upright in an anatomical position, by moving downwards at a constant speed over the SM spinal criterion points (from C7 spinous process to S3) by the physiotherapist. The spine is measured 3 times in the sagittal plane. The average value of the measurements is used for analysis.
Evaluation of Hand Functions | at baseline and week 9
  Jebsen Taylor Hand Function Test (JTHFT): Writing, card turning, picking up small objects, large and heavy objects skills and durations are assessed in both hands. 7 items are repeated for both hands. The completion time of each task is recorded separately. The score for the subtest is equal to the time in seconds required to complete the task, the maximum score for the subtest is 120. The total score is equal to the sum of points for all subtests and is calculated separately for each hand. The lower the score, the better the child's hand function.

SECONDARY OUTCOMES:
1 Minute Walking Test (1-MWT): | at baseline and week 9
  The 1-minute walk test (1-MWT) is a valid and simple assessment for monitoring changes in walking capacity in children with chronic conditions. While performing the 1-MWT, children are asked to walk as fast as they can on a circular track. Running is prohibited. They may use mobility aids if necessary. The distance they travel on the track is recorded.
Pediatric Data Collection Tool (PODCI) | at baseline and week 9
  PODCI consists of 5 subscales: Upper Extremity and Physical Function, Transfer and Basic Mobility, Pain/Comfort, Happiness, Sports and Physical Function, and Global Function. PODCI scores are calculated separately for each subscale and range from 0 to 100 points. Higher scores represent better health. The PODCI includes 86 items in 3 scales: global function, happiness, and expectations. The global function scale is the average of 4 subscales: upper extremity and physical function, transfers and basic mobility, sports and physical function, and pain and comfort. Items are scored ranging from 0 to 3 and 0 to 6, with lower scores indicating higher disability level.

CONTACTS AND LOCATIONS:
Overall Officials: Seval KUTLUTÜRK YIKILMAZ, PhD, Principal Investigator — University of Health Sciences Hamidiye Faculty of Health Sciences; Orçun TOKTAŞ, Op. Dr, Principal Investigator — Etimesgut Şehit Sait Ertürk State Hospital Orthopedics and Traumatology.; Gül EVDALI, MScPT, Principal Investigator — University of Health Sciences Hamidiye Health Sciences Institute
Locations (3):
- Turkey (Türkiye) (3):
  - Sacettin Gürbüz Barrier-Free Life Center (General name of the campus.) /*Private Etimesgut Barrier-Free Life Special Education and Rehabilitation Center, Ankara, Etimesgut
  - Private Etimesgut Kardelen Special Education and Rehabilitation Center, Ankara, Etimesgut
  - SERÇEV Barrier-Free and Vocational Technical Anatolian High School, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Giannoni P, Zerbino L. Cerebral Palsy: A Practical Guide for Rehabilitation Professionals. Springer International Publishing; 2022. https://books.google.com.tr/books?id=apxhEAAAQBAJ
- [Background] Dewar R, Love S, Johnston LM. Exercise interventions improve postural control in children with cerebral palsy: a systematic review. Dev Med Child Neurol. 2015 Jun;57(6):504-20. doi: 10.1111/dmcn.12660. Epub 2014 Dec 18. PMID 25523410
- [Background] 3. Akbaş AN, Günel MK. Effects of individually structured trunk training on body function and structures in children with spastic cerebral palsy: A stratified randomized controlled trial. In: Turkish Journal of Physiotherapy and Rehabilitation. Turkish Physiotherapy Association; 2019;30(1) 11-22.
- [Background] Ruthard K, Raabe-Oetker A, Ruthard J, Oppermann T, Duran I, Schonau E. Reliability of a radiation-free, noninvasive and computer-assisted assessment of the spine in children with cerebral palsy. Eur Spine J. 2020 May;29(5):937-942. doi: 10.1007/s00586-020-06328-4. Epub 2020 Feb 8. PMID 32036426
- [Background] Pierret J, Beyaert C, Vasa R, Rumilly E, Paysant J, Caudron S. Rehabilitation of Postural Control and Gait in Children with Cerebral Palsy: the Beneficial Effects of Trunk-Focused Postural Activities. Dev Neurorehabil. 2023 Apr;26(3):180-192. doi: 10.1080/17518423.2023.2193269. Epub 2023 Mar 23. PMID 36959769
- [Background] Talgeri AJ, Nayak A, Karnad SD, Jain P, Tedla JS, Reddy RS, Sangadala DR. Effect of Trunk Targeted Interventions on Functional Outcomes in Children with Cerebral Palsy- A Systematic Review. Dev Neurorehabil. 2023 Apr;26(3):193-205. doi: 10.1080/17518423.2023.2193265. Epub 2023 Apr 5. PMID 37021364
- [Background] Faccioli S, Pagliano E, Ferrari A, Maghini C, Siani MF, Sgherri G, Cappetta G, Borelli G, Farella GM, Foscan M, Vigano M, Sghedoni S, Perazza S, Sassi S. Evidence-based management and motor rehabilitation of cerebral palsy children and adolescents: a systematic review. Front Neurol. 2023 May 25;14:1171224. doi: 10.3389/fneur.2023.1171224. eCollection 2023. PMID 37305763
- [Background] 8. Kisner, C., Colby, L. A., Borstad, J. (2022). Therapeutic Exercise: Foundations and Techniques. United States: F.A. Davis.
- [Background] Monticone M, Ambrosini E, Cazzaniga D, Rocca B, Ferrante S. Active self-correction and task-oriented exercises reduce spinal deformity and improve quality of life in subjects with mild adolescent idiopathic scoliosis. Results of a randomised controlled trial. Eur Spine J. 2014 Jun;23(6):1204-14. doi: 10.1007/s00586-014-3241-y. Epub 2014 Feb 28. PMID 24682356
- [Background] 11. Martin, S. C.(2018). Spinal Asymmetry and Scoliosis: Movement and Function Solutions for the Spine, Ribcage and Pelvis. p. 213. Jessica Kingsley Publishers.
- [Background] 15. Mendoza, A. et all. (Ed) (2023, July 20).
- [Background] 13. Lenhert-Schroth, C. (2007). The Schroth scoliosis three dimensional treatment. Books on Demand GmbH. https://books.google.com.tr/books?id=D0gQAQAAMAAJ&dq=9780914959021,&hl=en&newbks=1&newbks_redir=1&sa=X&ved=2ahUKEwibwbfyp82JAxV_RfEDHZbSG3IQ6AF6BAgGEAI
- See also: 1. Giannoni, P., & Zerbino, L. (2022). Cerebral Palsy: A Practical Guide for Rehabilitation Professionals. In Google Books. Springer Nature. https://books.google.com.tr/books?id=apxhEAAAQBAJ — https://books.google.com.tr/books?id=apxhEAAAQBAJ
- See also: 2. Dewar, R., Love, S., & Johnston, L. M. (2015). Exercise interventions improve postural control in children with cerebral palsy: a systematic review. Developmental medicine and child neurology, 57(6), 504-520. https://doi.org/10.1111/dmcn.12660 — https://pubmed.ncbi.nlm.nih.gov/25523410/
- See also: 3. Numanoğlu Akbaş, A., & Kerem Günel, M. (2019). EFFECTS OF INDIVIDUALLY STRUCTURED TRUNK TRAINING ON BODY FUNCTION AND STRUCTURES IN CHILDREN WITH SPASTIC CEREBRAL PALSY: A STRATIFIED RANDOMIZED CONTROLLED TRIAL. Fizyoterapi Rehabilitasyon, 30(1),11-22 — https://dergipark.org.tr/tr/pub/tfrd/issue/45078/382366
- See also: 4. Ruthard, Kristina et al. "Reliability of a radiation-free, noninvasive and computer-assisted assessment of the spine in children with cerebral palsy." European spine journal : official publication of the European Spine Society. — https://pubmed.ncbi.nlm.nih.gov/32036426/
- See also: 5. Pierret, Jonathan et al. "Rehabilitation of Postural Control and Gait in Children with Cerebral Palsy: the Beneficial Effects of Trunk-Focused Postural Activities." Developmental neurorehabilitation vol. 26,3 (2023): 180-192. doi:10.1080/17518423.2023 — https://pubmed.ncbi.nlm.nih.gov/36959769/
- See also: 6. Faccioli, S., Pagliano, E., Ferrari, A., Maghini, C., Siani, M. F., Sgherri, G., Cappetta, G., Borelli, G., Farella, G. M., Foscan, M., Viganò, M., Sghedoni, S., Perazza, S., & Sassi, S. (2023). Evidence-based management and motor rehabilitation of ce — https://pubmed.ncbi.nlm.nih.gov/37305763/
- See also: 7. Talgeri, A. J., Nayak, A., Karnad, S. D., Jain, P., Tedla, J. S., Reddy, R. S., & Sangadala, D. R. (2023). Effect of Trunk Targeted Interventions on Functional Outcomes in Children with Cerebral Palsy- A Systematic Review. Developmental neurorehabilit — https://pubmed.ncbi.nlm.nih.gov/37021364/
- See also: 8. Kisner, C., Colby, L. A., & Borstad, J. (2022). Therapeutic Exercise : Foundations and Techniques. In Google Books. F.A. Davis. https://books.google.com.tr/books?id=xKegEAAAQBAJ — https://books.google.com.tr/books?id=xKegEAAAQBAJ
- See also: 9. Schroth, C. L. (2007). Three-Dimensional Treatment for scoliosis: a physiotherapeutic method for deformities of the spine: 9780914959021: Medicine & Health Science Books @ Amazon.com (C. Mohr, A. Reeves, & D. A. Smith, Trans.; 1st English edition). Th — https://www.amazon.com/Three-Dimensional-Treatment-Scoliosis-Physiotherapeutic-Deformities/dp/0914959026
- See also: 10. Kuru Çolak, T., Akçay, B., & Apti, A. (2020). Skolyoz Tedavisinde Schroth Yöntemi. Hacettepe University Faculty of Health Sciences Journal, 7(1), 1-12. https://doi.org/10.21020/husbfd.601264 — https://doi.org/10.21020/husbfd.601264
- See also: 11. Esquerdo, O. M. (2016). Stretching Exercises Encyclopedia. In Google Books: Vol. p. 52 (illustrated ed.). Meyer & Meyer Verlag. https://books.google.com.tr/books?id=3-TvkJgmE6cC&source=gbs_navlinks_s — https://books.google.com.tr/books?id=3-TvkJgmE6cC&source=gbs_navlinks_s
- See also: 12. Monticone, M., Ambrosini, E., Cazzaniga, D., Rocca, B., & Ferrante, S. (2014). Active self-correction and task-oriented exercises reduce spinal deformity and improve quality of life in subjects with mild adolescent idiopathic scoliosis. Results of a — https://pubmed.ncbi.nlm.nih.gov/24682356/
- See also: 13. Kotwicki, T., & Grivas, T. B. (2012). Research into spinal deformities 8. — https://search.library.ucsf.edu/permalink/01UCS_SAF/88i771/alma991000017589706536
- See also: 14. Martin, S. C. (2018). Spinal Asymmetry and Scoliosis: movement and function solutions for the spine, ribcage and pelvis. In Google Books: Vol. p.213 (illustrated ed.). Jessica Kingsley Publishers. https://books.google.com.tr/books?id=hJhsvgAACAAJ — https://books.google.com.tr/books?id=hJhsvgAACAAJ
- See also: 15. Mendoza et all, 2023, para.1-4. — https://www.scribd.com/document/742070779/The-ScoliClinic-5-Tips-For-Supporting-Your-Scoliosis-While-You-Sleep
- See also: 16. Monroe, M. (2012). Yoga and Scoliosis: A Journey to Health and Healing (16pt Large Print Edition). ReadHowYouWant. — https://www.google.com.tr/books/edition/Yoga_and_Scoliosis/qaJrmefYYcwC?hl=tr&gbpv=1&dq=good%20sitting%20scoliosis&pg=PA237&printsec=frontcover
- See also: 17. Krentzman, R. (2016). Scoliosis, Yoga Therapy, and the Art of Letting Go. Birleşik Krallık: Jessica Kingsley Publishers.p.53-57 — https://www.google.com.tr/books/edition/Scoliosis_Yoga_Therapy_and_the_Art_of_Le/DuXiDAAAQBAJ?hl=en&gbpv=0
- Available data/document: Statistical Analysis Plan: gulevdali@hotmail.com — https://www.akademikredaksiyon.com/ — The study data is shared with the official at the website https://www.akademikredaksiyon.com/ for statistical analysis and evaluation of the results.